CLINICAL TRIAL: NCT01311258
Title: A Program for Monitoring Minimal Residual Disease Following Treatment of Patients With Acute Myeloid Leukemia or High Grade Myelodysplastic Syndrome
Brief Title: Monitoring Minimal Residual Disease of Patients With Acute Myelogenous Leukemia or High Grade Myelodysplastic Syndrome
Acronym: MRD
Status: Recruiting | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Jane Liesveld, Principal Investigator, University of Rochester
Other Study IDs: 20123
Record Dates: First submitted 2011-03-07; First posted 2011-03-09 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood and bone marrow aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is being performed to develop assays to determine the impact of the therapy patients receive for treatment of AML or MDS and to determine if these tests can identify those patients who are at a greater risk for having their disease relapse.

DETAILED DESCRIPTION:
Following therapy, the majority of patients with AML and many patients with MDS will achieve a remission that is defined by the lack of any evidence of the disease when viewing bone marrow samples under a microscope. Despite the absence of disease by this method, many patients in remission will still have what is referred to as Minimal Residual Disease when more sensitive methods are applied. The presence of Minimal Residual Disease following therapy does not guarantee that the patient will experience a relapse. This is likely a result of the failure of these techniques to examine those cells that are responsible for disease relapse. Recent data suggests that in the majority of patients with AML or MDS only a minor population of the malignant cells are capable of maintaining the disease and are likely responsible for relapse following therapy. This minor population of cells can be identified by the proteins they have on their surface. This study tests the ability to identify Minimal Residual Disease following therapy by performing special assays that specifically target this minor population of malignant cells.

ELIGIBILITY:
Inclusion Criteria:

* Are being evaluated for the diagnosis and/or treatment of Acute Myelogenous Leukemia or High Grade myelodysplastic syndrome (defined as greater than 10 percent blasts on examination of the bone marrow aspirate).
* Have not undergone prior cytotoxic therapy for acute myelogenous leukemia or High Grade myelodysplastic syndrome in the past 3 months other than hydroxyurea or Revlimid.
* Have not previously received an allogeneic peripheral blood or bone marrow stem cell transplant for their disease.
* Are able to sign an informed consent. Informed consent must be signed at the time of enrollment and prior to the collection of any specimens and/or clinical data (other than PHI needed to screen and identify patients, which will be promptly discarded in a secure fashion if patient is not enrolled on study)
* Are at least 18 years of age.
* Do not have any serious medical or psychiatric illness, other than that treated by this study which would limit the ability of the patient to receive therapy or give informed consent.
* Have been informed of the investigational nature of this study and given written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Subjects who are less than 18 years of age.
* Subjects with limited decision making capacity.
* Subjects who have received prior cytotoxic therapy, other than hydroxyurea or Revlimid, for their disease within the past three months.
* Patients with a diagnosis of chronic myelogenous leukemia in blast crisis, Acute Promyelocytic Leukemia, or Bi-lineage leukemia.
* Subjects who have previously undergone an allogeneic peripheral blood stem cell transplant.
* Have an active malignancy other than acute myelogenous leukemia (AML) or myelodysplastic syndrome (MDS) at the time of evaluation or a prior history of treatment for a malignancy other than AML or MDS within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematology/oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-08; Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Identification of Minimal Residual Disease after treatment for disease | 2 years
  To test the ability to identify Minimal Residual Disease following therapy by performing special assays that specifically target this minor population of malignant cells by evaluating the expression of cell surface antigens previously shown to be informative.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Becker, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States